CLINICAL TRIAL: NCT05063773
Title: Novel Wireless Mixed Reality Headset for Image Guidance in Cardiac Catheterization Laboratory
Acronym: MRCCL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SG Devices LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUD_002
Record Dates: First submitted 2021-09-08; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Radiation Injuries
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Device: Mixed reality heads up display
- Group 2 (No Intervention)

INTERVENTIONS:
Device: Mixed reality heads up display — Physician will use a mixed reality headset for image guidance of the procedure
  Arms: Group 1

SUMMARY:
Our hypothesis is that improved line of sight to patient data, ergonomics, and headset lead shielding in the CCL will lead to behavioral changes in the CCL personnel that will reduce radiation exposure to all members of the team. Further, reducing the burden of large, cumbersome monitors will enable improved use of shielding. Our approach is a single center randomized controlled trial of consecutive patients randomly assigned to one of two groups with group 1 using mixed reality display and group 2 using standard 2D displays to perform diagnostic angiography in the CCL. Radiation exposure will be evaluated at multiple levels including total radiation exposure, exposure of each individual staff member, as well as specific exposure to eyes and head in group 1 versus group 2.

ELIGIBILITY:
Inclusion Criteria:

* undergoing diagnostic coronary angiography

Exclusion Criteria:

* acute coronary syndrome, cardiogenic shock, cardiac arrest, planned intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Radiation exposure to the physician | up to 24 months

SECONDARY OUTCOMES:
radiation exposure to the patient and medical staff | up to 24 months

IPD SHARING:
Plan to Share IPD: No